CLINICAL TRIAL: NCT01493973
Title: A Double-blind, Randomized, Placebo-controlled, Clinical Trial to Test the Efficacy of Epoetin Alfa on Physical Performance of Friedreich Ataxia Patients.
Brief Title: Efficacy Study of Epoetin Alfa in Friedreich Ataxia
Acronym: FRIEMAX
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Federico II University (Other)
Collaborators: Friedreich's Ataxia Research Alliance (Other); Associazione Italiana per la lotta alle Sindromi Atassiche (AISA) (Unknown)
Responsible Party: Principal Investigator, Alessandro Filla, Principal Investigator, Federico II University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FA_BBK_8
Record Dates: First submitted 2011-12-15; First posted 2011-12-16 (Estimated); Last update posted 2015-08-11 (Estimated); Status verified 2015-08

CONDITIONS: Friedreich Ataxia
Keywords: Erythropoietin; EPO; Friedreich; Ataxia; Epoetin alfa; VO2 max; SARA; EQ-5D; frataxin
MeSH Terms: conditions — Friedreich Ataxia; Ataxia | interventions — Epoetin Alfa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Epoetin alfa (Experimental): Patients will be treated with Epoetin alfa 1200 IU/Kg s.c. every 12 weeks
  Interventions: Drug: Epoetin alfa
- Placebo (Placebo Comparator): Placebo 1200 IU/Kg s.c. every 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Epoetin alfa — Epoetin alfa will be administered s.c. at 1200 IU/Kg every 12 weeks
  Other Names: EPREX 40000 IU; EPREX 10000 IU
  Arms: Epoetin alfa
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Friedreich's ataxia (FRDA) is a rare genetic disorder characterised by severe neurological disability and cardiomyopathy. Friedreich's ataxia is the consequence of frataxin deficiency. Although several drugs have been proposed, there is no available treatment. Four trials recently demonstrated that erythropoietin can increase the intracellular levels of frataxin. The present project is aimed at testing a long term therapeutic approach using erythropoietin, which is an already available and commercialised drug. The study will test the effect of erythropoietin on exercise capacity, which is reduced in patients with FRDA. Additional objectives of the study will be the drug's safety and tolerability, and its effect on frataxin, blood vessel reactivity, heart functional indexes, and disease progression.

DETAILED DESCRIPTION:
Friedreich's ataxia (FA) is an autosomal recessive ataxia caused by a trinucleotide GAA expansion in the first intron of the FXN gene. The gene encodes for a 210aa mitochondrial protein called frataxin, whose mRNA and protein levels are severely reduced in FA. It has been suggested that frataxin is involved in iron-sulphur cluster and heme biogenesis, iron binding/storage, and chaperone activity. Clinically, the age of onset is generally around puberty and, as the disease progresses, there is increasing ataxia of the limbs, and eventually most patients are wheelchair bound by the twenties. Cardiomyopathy with myocardial hypertrophy occurs very often and is the predominant cause of death. Type II diabetes, scoliosis, foot deformities, optic atrophy, and deafness are other relatively frequent symptoms.

Erythropoietin (EPO) is a glycoprotein that acts as a main regulator for erythropoiesis. Evidence suggests that both EPO and its receptor are expressed in the nervous tissue, and neuroprotective effects have been shown in animal models of cerebral ischemic damage. EPO increases frataxin levels in cultured human lymphocytes from FRDA patients. However, frataxin protein increase is not preceded by mRNA increase, suggesting that a post-transcriptional mechanism is involved. To date, four phase II clinical trials have been published regarding the use of EPO in FRDA patients.

ELIGIBILITY:
Inclusion Criteria:

* Molecular diagnosis of Friedreich Ataxia
* Age ≥12 years
* Body weight ≥30, ≤90 Kg
* SARA score ≤30
* Patient able to read and sign the informed consent
* Patients able to perform a cardiopulmonary test

Exclusion Criteria:

* Treatment with Erythropoietin in the previous 12 months
* Treatment with Idebenone
* Contraindications to CPET: cardiac valve disease, ischemic cardiomyopathy, atrial fibrillation, asthma, chronic obstructive pulmonary disease, other arrhythmias judged as not compatible with exercise.
* Any Cardiac and/or Hepatic and/or Renal disease judged as clinically relevant by the investigator
* Any clinically relevant ECG abnormalities that may interfere with the study
* Any abnormal and clinically relevant laboratory exams at screening visit that may interfere with the trial
* Anemia with Hemoglobin <10 g/dL
* Positive history for venous and/or arterial thrombosis
* Drug-resistant arterial hypertension
* Positive history for drug-resistant epilepsy
* Patients in treatment with not allowed study drugs (starting from 3 months prior to screening)
* Any acute/chronic disease that might interfere with the clinical trial, as judged by the investigator
* Hypersensitivity to Epoetin alfa or any other component of the study drug
* Patients not able to comply to the study
* For female patients (Sexually not active, hysterectomized, sterilized, menopause patients are excluded from the following criteria): pregnancy and/or breastfeeding and/or inadequate contraception.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2013-01; Primary Completion 2014-10 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Peak oxygen uptake (VO2 max) at the cardiopulmonary exercise test (CPET) | 48 weeks
  Patients will undergo a complete CPET as described in the methods section. CPET will be performed at baseline (Visit 2), at 24 weeks (Visit 5), and at 48 weeks (Visit 7).

SECONDARY OUTCOMES:
Secondary outcome variables at the CPET (anaerobic threshold, ventilatory efficiency, exercise duration, and power output). | 24 and 48 weeks
Frataxin levels in peripheral blood mononuclear cells (PBMCs). | all timepoints
Echocardiography | 24, and 48 weeks
Vascular reactivity | 24 and 48 weeks
  Vascular reactivity will be measured by the Flow-Mediated Dilation technique (FMD)
Neurological progression | 24 and 48 weeks
  Neurological progression will be measured with the Scale for the Assessment and Rating of Ataxia (SARA), and with the 9 hole pegboard test (9-HPT)
Quality of life | 24 and 48 weeks
  Quality of life will be assessed with the EQ-5D, ADL, and IADL scales
Safety and tolerability | all visits
  Safety and tolerability will be assessed by recording all serious and non serious adverse events at all visits of the trial

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Saccà, MD, Study Director — University Federico II, Naples Italy
Locations (3):
- Italy (3):
  - Università di Bari, Bari, BA
  - Università la Sapienza, Neurologia C, Rome, RM
  - Dipartimento di Scienze Neurologiche, Napoli

REFERENCES:
- [Background] Sacca F, Piro R, De Michele G, Acquaviva F, Antenora A, Carlomagno G, Cocozza S, Denaro A, Guacci A, Marsili A, Perrotta G, Puorro G, Cittadini A, Filla A. Epoetin alfa increases frataxin production in Friedreich's ataxia without affecting hematocrit. Mov Disord. 2011 Mar;26(4):739-42. doi: 10.1002/mds.23435. Epub 2010 Nov 10. PMID 21506154
- [Background] Acquaviva F, Castaldo I, Filla A, Giacchetti M, Marmolino D, Monticelli A, Pinelli M, Sacca F, Cocozza S. Recombinant human erythropoietin increases frataxin protein expression without increasing mRNA expression. Cerebellum. 2008;7(3):360-5. doi: 10.1007/s12311-008-0036-x. PMID 18581197
- [Background] Boesch S, Sturm B, Hering S, Scheiber-Mojdehkar B, Steinkellner H, Goldenberg H, Poewe W. Neurological effects of recombinant human erythropoietin in Friedreich's ataxia: a clinical pilot trial. Mov Disord. 2008 Oct 15;23(13):1940-4. doi: 10.1002/mds.22294. PMID 18759345
- [Background] Boesch S, Sturm B, Hering S, Goldenberg H, Poewe W, Scheiber-Mojdehkar B. Friedreich's ataxia: clinical pilot trial with recombinant human erythropoietin. Ann Neurol. 2007 Nov;62(5):521-4. doi: 10.1002/ana.21177. PMID 17702040
- [Background] Sturm B, Stupphann D, Kaun C, Boesch S, Schranzhofer M, Wojta J, Goldenberg H, Scheiber-Mojdehkar B. Recombinant human erythropoietin: effects on frataxin expression in vitro. Eur J Clin Invest. 2005 Nov;35(11):711-7. doi: 10.1111/j.1365-2362.2005.01568.x. PMID 16269021
- See also: Clinical trials site — http://www.neurologia.unina.it
- See also: University Federico II, Naples Italy — http://www.unina.it
- See also: Friedreich Ataxia Research Alliance — http://www.curefa.org
- See also: Associazione Italiana per la lotta alle Sindromi Atassiche — http://www.atassia.it